CLINICAL TRIAL: NCT01369342
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study to Evaluate the Safety and Efficacy of Ustekinumab Induction Therapy in Subjects With Moderately to Severely Active Crohn's Disease (UNITI-2)
Brief Title: A Study to Evaluate the Safety and Efficacy of Ustekinumab Induction Therapy in Patients With Moderately to Severely Active Crohn's Disease (UNITI-2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR018418; CNTO1275CRD3002 (Other: Janssen Research & Development, LLC); 2010-022759-42 (EudraCT Number)
Record Dates: First submitted 2011-06-07; First posted 2011-06-08 (Estimated); Results first posted 2017-01-06 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2016-11

CONDITIONS: Crohn's Disease; Inflammatory Bowel Disease; IBD; Colitis
Keywords: ustekinumab; moderately to severely active Crohn's Disease; Stelara; IBD; colitis; crohn; UNITI; Crohn's
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases; Colitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo IV (Placebo Comparator): Group 1: Placebo Form=solution for injection route=intravenous use in a single dose.
  Interventions: Drug: Group 1: Placebo
- Ustekinumab 130 milligram (mg) (Experimental): Group 2 ustekinumab 130 mg Type=exact unit=mg number=130 form=solution for injection route= intravenous use in a single dose.
  Interventions: Drug: Group 2 ustekinumab 130 mg
- Ustekinumab approximately (~) 6 milligram per kilogram (mg/kg) (Experimental): Group 3: ustekinumab approximately 6 mg/kg Type=range unit=mg/kg number=6 form=solution for injection route= intravenous use in a single dose.weight-range based ustekinumab doses approximating ustekinumab 6 mg/kg: 260 mg (weight <= 55 kg) 390 mg (weight > 55 kg and <= 85 kg) and 520 mg (weight > 85 kg).
  Interventions: Drug: Group 3: ustekinumab approximately 6 mg/kg

INTERVENTIONS:
Drug: Group 1: Placebo — Form=solution for injection, route=intravenous use, in a single dose.
  Arms: Placebo IV
Drug: Group 2 ustekinumab 130 mg — Type=exact, unit=mg, number=130, form=solution for injection, route= intravenous use, in a single dose.
  Arms: Ustekinumab 130 milligram (mg)
Drug: Group 3: ustekinumab approximately 6 mg/kg — Type=range, unit=mg/kg, number=6, form=solution for injection, route= intravenous use, in a single dose.weight-range based ustekinumab doses approximating ustekinumab 6 mg/kg: 260 mg (weight <= 55 kg), 390 mg (weight > 55 kg and <= 85 kg), and 520 mg (weight > 85 kg).
  Arms: Ustekinumab approximately (~) 6 milligram per kilogram (mg/kg)

SUMMARY:
This study (UNITI-2) will compare the effects (both positive and negative) of an initial treatment with ustekinumab to a placebo over 8 weeks in patients with moderately to severely active Crohn's disease.

DETAILED DESCRIPTION:
This study (CNTO1275CRD3002 or "UNITI-2") examines ustekinumab (an antibody medication that inhibits the inflammatory proteins IL-12 and IL-23) versus a placebo (otherwise identical except without the ustekinumab antibody) given intravenously (by an IV) in adults with moderately to severely active Crohn's disease. Ustekinumab (also known as Stelara) is approved as a treatment for the skin condition of moderate to severe plaque-type psoriasis, but this study will examine if ustekinumab can provide benefit in Crohn's disease and also assess for any risks or side effects. Both the positive and negative outcomes of IV placebo versus two different doses of IV ustekinumab will be tracked and compared over eight weeks, in approximately 612 patients who have previously failed or were intolerant to corticosteroids or immunomodulators (methotrexate, azathioprine, or 6-mercaptopurine) or are dependent on corticosteroid medications. Patients enrolling in this study will be assigned to one of the 3 treatment groups by chance (randomly, like rolling dice), and all will receive a single IV administration of study agent at the first study visit (after the screening period), and then will be asked to return for 3 additional visits through Week 8. Patients who complete this study through the Week 8 visit and remain eligible can enter the maintenance study (CNTO1275CRD3003 or "IM-UNITI"), where they will receive additional study agent, including the administration of ustekinumab in patients who receive placebo in this study and have not had improvement in their Crohn's disease. Patients who do not enter the CNTO1275CRD3003 study will have a final safety follow-up visit approximately 20 weeks after they received study agent when they entered into this study at the Week 0 visit. .All patients will receive a single intravenous (IV) administration of study drug (placebo or ustekinumab) at the start of the study.There are 3 treatment groups in this study: Group 1: Placebo; Group 2: ustekinumab 130 mg, Group 3: weight-range based ustekinumab doses approximating ustekinumab 6 mg/kg: 260 mg (weight <= 55 kg), 390 mg (weight > 55 kg and <= 85 kg), and 520 mg (weight > 85 kg).

ELIGIBILITY:
Inclusion Criteria:

* Have Crohn's disease of at least 3 months' duration with colitis, ileitis, or ileocolitis, confirmed at some time in the past by radiography, histology, or endoscopy
* Have active Crohn's disease, defined as a baseline Crohn Disease Activity Index (CDAI) score of >= 220 and <= 450, with confirmation of active inflammation
* Has failed conventional therapy as demonstrated by having received corticosteroids and/or immunomodulators(ie, AZA, MTX, or 6-MP) at adequate therapeutic doses OR Have a history of failure to respond to or tolerate an adequate course of corticosteroids and/or immunomodulators (ie, AZA, MTX, or 6-MP) at adequate therapeutic doses OR Is corticosteroid dependent or has had a history of corticosteroid dependency AND Has not previously demonstrated failure of or intolerance to 1 or more TNF-antagonist therapies (ie, infliximab, adalimumab, or certolizumab pegol) per study criteria
* Have screening laboratory test results within protocol-specified parameters

Exclusion Criteria:

* Patients who have had any kind of bowel resection within 6 months
* Are pregnant or planning pregnancy (both men and women) while enrolled in the study or for 20 weeks after receiving study agent
* Patients who have received infliximab, adalimumab or certolizumab pegol < = 8 weeks before the first administration of study drug
* Patients with certain complications of Crohn's disease that would make it hard to assess response to study drug
* Patients with a history of or ongoing chronic or recurrent infectious disease
* Patients who have previously received a biologic agent targeting IL-12 or IL-23, including but not limited to ustekinumab (CNTO 1275) or briakinumab (ABT-874)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Actual)
Dates: Start 2011-07; Primary Completion 2014-08 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (220):
- United States (84):
  - Tucson, Arizona
  - Little Rock, Arkansas
  - La Jolla, California
  - Los Angeles, California
  - San Diego, California
  - Santa Monica, California
  - Torrance, California
  - Lone Tree, Colorado
  - Boca Raton, Florida
  - Gainesville, Florida
  - Jacksonville, Florida
  - Largo, Florida
  - Miami, Florida
  - Naples, Florida
  - Port Orange, Florida
  - Winter Park, Florida
  - Athens, Georgia
  - Atlanta, Georgia
  - Decatur, Georgia
  - Macon, Georgia
  - Idaho Falls, Idaho
  - Chicago, Illinois
  - Clive, Iowa
  - Pratt, Kansas
  - Topeka, Kansas
  - Crestview Hills, Kentucky
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - Houma, Louisiana
  - New Orleans, Louisiana
  - Chevy Chase, Maryland
  - Columbia, Maryland
  - Towson, Maryland
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - Ann Arbor, Michigan
  - Chesterfield, Michigan
  - Novi, Michigan
  - Troy, Michigan
  - Ypsilanti, Michigan
  - Rochester, Minnesota
  - Jackson, Mississippi
  - Ocean Springs, Mississippi
  - Columbia, Missouri
  - Kansas City, Missouri
  - Lees Summit, Missouri
  - Urbana, Missouri
  - Las Vegas, Nevada
  - Egg Harbor, New Jersey
  - Marlton, New Jersey
  - Morristown, New Jersey
  - Great Neck, New York
  - New York, New York
  - Poughkeepsie, New York
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Raleigh, North Carolina
  - Beavercreek, Ohio
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Mentor, Ohio
  - Norman, Oklahoma
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Bend, Oregon
  - Portland, Oregon
  - Malvern, Pennsylvania
  - Philadelphia, Pennsylvania
  - Columbia, South Carolina
  - North Charleston, South Carolina
  - Germantown, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Grapevine, Texas
  - Houston, Texas
  - Tyler, Texas
  - Salt Lake City, Utah
  - Charlottesville, Virginia
  - Chesapeake, Virginia
  - Virginia Beach, Virginia
  - Bellevue, Washington
  - Seattle, Washington
  - Madison, Wisconsin
- Australia (9):
  - Adelaide
  - Cairns
  - Central Queensland M C
  - Concord
  - Fremantle
  - Garran
  - Liverpool
  - Malvern
  - Parkville
- Belgium (2):
  - Brussels
  - Leuven
- Brazil (4):
  - Goiânia
  - Porto Alegre
  - Rio de Janeiro
  - São Paulo
- Bulgaria (4):
  - Pleven
  - Rousse
  - Sofia
  - Varna
- Canada (11):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Brandon, Manitoba
  - Kingston, Ontario
  - London, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Saskatoon, Saskatchewan
  - Saskatoon
  - Winnipeg
- Croatia (3):
  - Osijek
  - Rijeka
  - Zagreb
- France (7):
  - Amiens
  - Bordeaux
  - Caen
  - Lille
  - Paris
  - Rouen
  - Vandœuvre-lès-Nancy
- Germany (17):
  - Berlin
  - Bochum
  - Frankfurt
  - Halle
  - Hamburg
  - Hanover
  - Haßloch
  - Heidelberg
  - Kiel
  - Lÿneburg
  - Mannheim
  - Minden
  - München
  - Münster
  - Regensburg
  - Stade
  - Ulm
- Hungary (8):
  - Békéscsaba
  - Budapest
  - Debrecen
  - Gyula
  - Mosonmagyaróvár
  - Pécs
  - Szekszárd
  - Székesfehérvár
- Reykjavik, Iceland
- Israel (7):
  - Beer Yaakov
  - Haifa
  - Jerusalem
  - Kfar Saba
  - Petah Tikva
  - Rehovot
  - Tel Aviv
- Japan (20):
  - Chikushino-shi
  - Hachiōji
  - Hamamatsu
  - Hirosaki
  - Hiroshima
  - Kagoshima
  - Nishinomiya
  - Ohtsu
  - Osaka
  - Ōita
  - Sakura
  - Sapporo
  - Sendai
  - Suita-Shi
  - Tokyo
  - Tsu
  - Uruma
  - Yokkaichi
  - Yokohama
  - Yokosuka
- Netherlands (4):
  - Amsterdam
  - Amsterdam-Zuidoost
  - Maastricht
  - Rotterdam
- New Zealand (8):
  - Auckland
  - Christchurch
  - Dunedin
  - Grafton
  - Hamilton
  - Hastings
  - Plenty
  - Wellington
- Poland (5):
  - Bydgoszcz
  - Elblag
  - Krakow
  - Lodz
  - Warsaw
- Russia (2):
  - Moscow
  - Novosibirsk
- Belgrade, Serbia
- South Africa (3):
  - Cape Town
  - Durban
  - Pretoria
- South Korea (3):
  - Daegu
  - Gyeonggi-do
  - Seoul
- Spain (3):
  - Madrid
  - Sabadell
  - Santiago de Compostela
- United Kingdom (14):
  - Birmingham
  - Brighton
  - Bristol
  - Cambridge
  - Gloucester
  - Harrow
  - Liverpool
  - London
  - Manchester
  - Norwich
  - Nottinghamshirecc
  - Oxford
  - Shrewsbury
  - Southampton

REFERENCES:
- [Derived] Ghosh S, Feagan BG, Ott E, Gasink C, Godwin B, Marano C, Miao Y, Ma T, Loftus EV Jr, Sandborn WJ, Danese S, Abreu MT, Sands BE. Safety of Ustekinumab in Inflammatory Bowel Disease: Pooled Safety Analysis Through 5 Years in Crohn's Disease and 4 Years in Ulcerative Colitis. J Crohns Colitis. 2024 Aug 6;18(7):1091-1101. doi: 10.1093/ecco-jcc/jjae013. PMID 38310565
- [Derived] Colombel JF, Sands BE, Gasink C, Yeager B, Adedokun OJ, Izanec J, Ma T, Gao LL, Lee SD, Targan SR, Ghosh S, Hanauer SB, Sandborn WJ. Evolution of Symptoms After Ustekinumab Induction Therapy in Patients With Crohn's Disease. Clin Gastroenterol Hepatol. 2024 Jan;22(1):144-153.e2. doi: 10.1016/j.cgh.2023.06.014. Epub 2023 Jun 28. PMID 37391056
- [Derived] Dubinsky M, Ma C, Griffith J, Crowell M, Neimark E, Kligys K, O'Connell T. Matching-Adjusted Indirect Comparison Between Risankizumab and Ustekinumab for Induction and Maintenance Treatment of Moderately to Severely Active Crohn's Disease. Adv Ther. 2023 Sep;40(9):3896-3911. doi: 10.1007/s12325-023-02546-6. Epub 2023 Jun 27. PMID 37368103
- [Derived] Adedokun OJ, Xu Z, Gasink C, Kowalski K, Sandborn WJ, Feagan B. Population Pharmacokinetics and Exposure-Response Analyses of Ustekinumab in Patients With Moderately to Severely Active Crohn's Disease. Clin Ther. 2022 Oct;44(10):1336-1355. doi: 10.1016/j.clinthera.2022.08.010. Epub 2022 Sep 21. PMID 36150926
- [Derived] Narula N, Aruljothy A, Wong ECL, Homenauth R, Alshahrani AA, Marshall JK, Reinisch W. The impact of ustekinumab on extraintestinal manifestations of Crohn's disease: A post hoc analysis of the UNITI studies. United European Gastroenterol J. 2021 Jun;9(5):581-589. doi: 10.1002/ueg2.12094. Epub 2021 Jun 2. PMID 34077627
- [Derived] Sandborn WJ, Feagan BG, Danese S, O'Brien CD, Ott E, Marano C, Baker T, Zhou Y, Volger S, Tikhonov I, Gasink C, Sands BE, Ghosh S. Safety of Ustekinumab in Inflammatory Bowel Disease: Pooled Safety Analysis of Results from Phase 2/3 Studies. Inflamm Bowel Dis. 2021 Jun 15;27(7):994-1007. doi: 10.1093/ibd/izaa236. PMID 32964215
- [Derived] Li K, Friedman JR, Chan D, Pollack P, Yang F, Jacobstein D, Brodmerkel C, Gasink C, Feagan BG, Sandborn WJ, Rutgeerts P, De Hertogh G. Effects of Ustekinumab on Histologic Disease Activity in Patients With Crohn's Disease. Gastroenterology. 2019 Oct;157(4):1019-1031.e7. doi: 10.1053/j.gastro.2019.06.037. Epub 2019 Jul 4. PMID 31279870
- [Derived] Ghosh S, Gensler LS, Yang Z, Gasink C, Chakravarty SD, Farahi K, Ramachandran P, Ott E, Strober BE. Ustekinumab Safety in Psoriasis, Psoriatic Arthritis, and Crohn's Disease: An Integrated Analysis of Phase II/III Clinical Development Programs. Drug Saf. 2019 Jun;42(6):751-768. doi: 10.1007/s40264-019-00797-3. PMID 30739254
- [Derived] Rutgeerts P, Gasink C, Chan D, Lang Y, Pollack P, Colombel JF, Wolf DC, Jacobstein D, Johanns J, Szapary P, Adedokun OJ, Feagan BG, Sandborn WJ. Efficacy of Ustekinumab for Inducing Endoscopic Healing in Patients With Crohn's Disease. Gastroenterology. 2018 Oct;155(4):1045-1058. doi: 10.1053/j.gastro.2018.06.035. Epub 2018 Aug 29. PMID 29909019
- [Derived] Adedokun OJ, Xu Z, Gasink C, Jacobstein D, Szapary P, Johanns J, Gao LL, Davis HM, Hanauer SB, Feagan BG, Ghosh S, Sandborn WJ. Pharmacokinetics and Exposure Response Relationships of Ustekinumab in Patients With Crohn's Disease. Gastroenterology. 2018 May;154(6):1660-1671. doi: 10.1053/j.gastro.2018.01.043. Epub 2018 Feb 1. PMID 29409871
- [Derived] Hibi T, Imai Y, Murata Y, Matsushima N, Zheng R, Gasink C. Efficacy and safety of ustekinumab in Japanese patients with moderately to severely active Crohn's disease: a subpopulation analysis of phase 3 induction and maintenance studies. Intest Res. 2017 Oct;15(4):475-486. doi: 10.5217/ir.2017.15.4.475. Epub 2017 Oct 23. PMID 29142515
- [Derived] Feagan BG, Sandborn WJ, Gasink C, Jacobstein D, Lang Y, Friedman JR, Blank MA, Johanns J, Gao LL, Miao Y, Adedokun OJ, Sands BE, Hanauer SB, Vermeire S, Targan S, Ghosh S, de Villiers WJ, Colombel JF, Tulassay Z, Seidler U, Salzberg BA, Desreumaux P, Lee SD, Loftus EV Jr, Dieleman LA, Katz S, Rutgeerts P; UNITI-IM-UNITI Study Group. Ustekinumab as Induction and Maintenance Therapy for Crohn's Disease. N Engl J Med. 2016 Nov 17;375(20):1946-1960. doi: 10.1056/NEJMoa1602773. PMID 27959607

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 640 participants were randomly assigned to receive study agent. The analyses (efficacy) were based on the 628 participants who were randomized after the study was restarted. However, one additional participant was excluded from efficacy analyses due to misconduct by the investigative site.
Pre-assignment Details: In November 2011, due to stability issue with the batch of the IV drug (130 mg Ustekinumab) sponsor temporarily suspended dosing of participants with ustekinumab. Study was restarted with 90 mg/ml on 17 February 2012.
Groups:
- Placebo IV: Participants randomized to receive a single dose of Placebo Intravenous (IV) infusion at week 0.
- Ustekinumab 130 Milligram (mg): Participants randomized to receive a single dose of ustekinumab 130 milligram (mg) IV at week 0.
- Ustekinumab Approximately (~) 6 Milligram Per Kilogram (mg/kg): Participants randomized to receive tiered ustekinumab dose approximately (~) 6 mg/kg IV at week 0. Ustekinumab 260 mg for participants body weight less than or equal to (< =) 55 kg, ustekinumab 390 mg for weight greater than (>) 55 kg and < = 85 kg and ustekinumab 520 mg for weight > 85 kg.
Period: Overall Study
Arm/Group | Placebo IV | Ustekinumab 130 Milligram (mg) | Ustekinumab Approximately (~) 6 Milligram Per Kilogram (mg/kg)
Started | 214 | 213 | 213
Completed | 201 | 204 | 210
Not Completed | 13 | 9 | 3
Not completed — Withdrawal by Subject | 7 | 7 | 2
Not completed — Lost to Follow-up | 5 | 2 | 1
Not completed — Not Treated | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo IV | Ustekinumab 130 Milligram (mg) | Ustekinumab Approximately (~) 6 Milligram Per Kilogram (mg/kg) | Total
Number analyzed (Participants) | 214 | 213 | 213 | 640
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (13.09) | 39.2 (13.74) | 38.8 (13.65) | 39.4 (13.48)
Gender [Count of Participants; unit: Participants]
  Female | 113 | 107 | 122 | 342
  Male | 101 | 106 | 91 | 298
Region of Enrollment [Number; unit: participants]
  Australia | 8 | 7 | 5 | 20
  Belgium | 1 | 1 | 2 | 4
  Bulgaria | 8 | 5 | 11 | 24
  Brazil | 2 | 5 | 2 | 9
  Canada | 14 | 18 | 10 | 42
  Germany | 19 | 15 | 13 | 47
  Spain | 0 | 1 | 0 | 1
  France | 3 | 2 | 5 | 10
  United Kingdom | 8 | 8 | 5 | 21
  Croatia | 1 | 2 | 1 | 4
  Hungary | 23 | 20 | 18 | 61
  Iceland | 0 | 1 | 1 | 2
  Israel | 2 | 3 | 6 | 11
  Italy | 2 | 2 | 5 | 9
  Japan | 9 | 8 | 9 | 26
  Korea | 7 | 7 | 6 | 20
  Netherland | 1 | 1 | 2 | 4
  New Zealand | 2 | 8 | 4 | 14
  Poland | 8 | 8 | 10 | 26
  Russia | 6 | 6 | 5 | 17
  Serbia | 4 | 8 | 3 | 15
  United States | 72 | 72 | 76 | 220
  South Africa | 14 | 5 | 14 | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Response at Week 6
Description: Clinical response at Week 6 was defined as a reduction from baseline in the Crohn's Disease Activity Index (CDAI) score of greater than or equal (>=) 100 points (in general, CDAI score ranges from 0 to approximately 600; higher score indicates higher disease activities). Participants with a baseline CDAI score of > = 220 to less than or equal (< =) 248 were considered to be in clinical response if a CDAI score of less than (<) 150 was attained. A decrease in CDAI score over time indicates improvement in disease activity.
Time Frame: Week 6
Population: Efficacy analyses set included all the participants who were randomized after the study was restarted.
Measure: Number; unit: participants
Groups:
- Placebo: Participants randomized to receive a single dose of Placebo Intravenous (IV) infusion at week 0.
- Ustekinumab 130 mg: Participants randomized to receive a single dose of ustekinumab 130 milligram (mg) IV at week 0.
Arm/Group | Placebo | Ustekinumab 130 mg | Ustekinumab Approximately (~) 6 Milligram Per Kilogram (mg/kg)
Number analyzed (Participants) | 209 | 209 | 209
participants | 60 | 108 | 116
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab 130 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test — A fixed sequence testing procedure was used to control alpha at 0.05 over the outcome measures; 2-sided Cochran-Mantel-Haenszel chi-square test, stratified by study region (Asia, Eastern Europe, or rest of world) and CDAI score (=< 300 or >300)
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab Approximately (~) 6 Milligram Per Kilogram (mg/kg); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test — A fixed sequence testing procedure was used to control alpha at 0.05 over the outcome measures; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: Number of Participants in Clinical Remission at Week 8
Description: Clinical remission at Week 8 was defined as a Crohn's Disease Activity Index (CDAI) score of <150 points.
Time Frame: Week 8
Population: Efficacy analyses set included all the participants who were randomized after the study was restarted.
Measure: Number; unit: participants
Arm/Group | Placebo | Ustekinumab 130 mg | Ustekinumab Approximately (~) 6 Milligram Per Kilogram (mg/kg)
Number analyzed (Participants) | 209 | 209 | 209
participants | 41 | 64 | 84
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab 130 mg; Test type: Superiority or Other; p = 0.009, Cochran-Mantel-Haenszel chi-square test — A fixed sequence testing procedure was used to control alpha at 0.05 over the outcome measures; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab Approximately (~) 6 Milligram Per Kilogram (mg/kg); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test — A fixed sequence testing procedure was used to control alpha at 0.05 over the outcome measures; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Participants in Clinical Response at Week 8
Description: Clinical response at Week 8 was defined as a reduction from baseline in the CDAI score of greater than or equal (>=) 100 points (in general, CDAI score ranges from 0 to approximately 600; higher score indicates higher disease activities). Participants with a baseline CDAI score of > = 220 to less than or equal (< =) 248 were considered to be in clinical response if a CDAI score of less than (<) 150 was attained. A decrease in CDAI score over time indicates improvement in disease activity.
Time Frame: Week 8
Population: Efficacy analyses set included all the participants who were randomized after the study was restarted.
Measure: Number; unit: participants
Arm/Group | Placebo | Ustekinumab 130 mg | Ustekinumab Approximately (~) 6 Milligram Per Kilogram (mg/kg)
Number analyzed (Participants) | 209 | 209 | 209
participants | 67 | 99 | 121
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab 130 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test — A fixed sequence testing procedure was used to control alpha at 0.05 over the outcome measures; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab Approximately (~) 6 Milligram Per Kilogram (mg/kg); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test — A fixed sequence testing procedure was used to control alpha at 0.05 over the outcome measures; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Number of Participants With Crohn's Disease Activity Index (CDAI) 70 Point Response at Week 6
Description: 70-point response is defined as at least 70 points reduction in CDAI score (in general, CDAI score ranges from 0 to approximately 600; higher score indicates higher disease activities). The CDAI score is used to quantify the symptoms of participants with Crohn's Disease. A decrease in CDAI over time indicates improvement in disease activity.
Time Frame: Week 6
Population: Efficacy analyses set included all the participants who were randomized after the study was restarted.
Measure: Number; unit: participants
Arm/Group | Placebo | Ustekinumab 130 mg | Ustekinumab Approximately (~) 6 Milligram Per Kilogram (mg/kg)
Number analyzed (Participants) | 209 | 209 | 209
participants | 81 | 123 | 135
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab 130 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test — A fixed sequence testing procedure was used to control alpha at 0.05 over the outcome measures; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab Approximately (~) 6 Milligram Per Kilogram (mg/kg); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test — A fixed sequence testing procedure was used to control alpha at 0.05 over the outcome measures; [statistical method as in outcome 1, analysis 1]

5. Secondary Outcome: Number of Participants With CDAI 70 Point Response at Week 3
Description: as for outcome 4
Time Frame: Week 3
Population: Efficacy analyses set included all the participants who were randomized after the study was restarted.
Measure: Number; unit: participants
Arm/Group | Placebo | Ustekinumab 130 mg | Ustekinumab Approximately (~) 6 Milligram Per Kilogram (mg/kg)
Number analyzed (Participants) | 209 | 209 | 209
participants | 66 | 103 | 106
Statistical Analysis 1: Comparison: Placebo vs Ustekinumab 130 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test — A fixed sequence testing procedure was used to control alpha at 0.05 over the outcome measures; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Ustekinumab Approximately (~) 6 Milligram Per Kilogram (mg/kg); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel chi-square test — A fixed sequence testing procedure was used to control alpha at 0.05 over the outcome measures; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to Week 8 for all participants (for participants who do not enter the maintenance study, adverse events will be collected up to 20 weeks after the study agent administration)
Description: 1 participant randomized to placebo never received study agent (not included in the AE analysis) and 1 participant randomized to placebo received ustekinumab (analyzed for safety in 130 mg group);2 participants randomized to -6 mg/kg received dose closer to 130 mg of ustekinumab (analyzed for safety in 130 mg group).
Groups:
- Placebo IV: Participants received single dose of Placebo Intravenous (IV) infusion at week 0.
- Ustekinumab 130 Milligram (mg): Participants received single dose of ustekinumab 130 milligram (mg) IV at week 0.
- Ustekinumab Approximately (~) 6 Milligram Per Kilogram (mg/kg): Participants received a single tiered ustekinumab dose approximately (~) 6 mg/kg IV at week 0. Ustekinumab 260 mg for participants body weight less than or equal to (< =) 55 kg, ustekinumab 390 mg for weight greater than (>) 55 kg and < = 85 kg and ustekinumab 520 mg for weight > 85 kg.
Arm/Group | Placebo IV | Ustekinumab 130 Milligram (mg) | Ustekinumab Approximately (~) 6 Milligram Per Kilogram (mg/kg)
Serious Adverse Events (participants affected / at risk) | 15/212 | 10/216 | 9/211
Other Adverse Events (participants affected / at risk) | 44/212 | 40/216 | 44/211
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo IV (N=212) | Ustekinumab 130 Milligram (mg) (N=216) | Ustekinumab Approximately (~) 6 Milligram Per Kilogram (mg/kg) (N=211)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Crohn's Disease (Gastrointestinal disorders) | 5 | 5 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Localised Intraabdominal Fluid Collection (Gastrointestinal disorders) | 0 | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 1 | 2
Small Intestinal Perforation (Gastrointestinal disorders) | 1 | 0 | 0
Chest Pain (General disorders) | 0 | 0 | 1
Impaired Healing (General disorders) | 0 | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 1 | 0
Bile Duct Stone (Hepatobiliary disorders) | 1 | 0 | 0
Anal Abscess (Infections and infestations) | 3 | 2 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Genital Herpes (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Incisional Hernia (Injury, poisoning and procedural complications) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0
Pneumothorax Spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary Granuloma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo IV (N=212) | Ustekinumab 130 Milligram (mg) (N=216) | Ustekinumab Approximately (~) 6 Milligram Per Kilogram (mg/kg) (N=211)
Nausea (Gastrointestinal disorders) | 5 | 7 | 11
Pyrexia (General disorders) | 10 | 6 | 11
Nasopharyngitis (Infections and infestations) | 10 | 10 | 14
Upper Respiratory Tract Infection (Infections and infestations) | 11 | 4 | 7
Headache (Nervous system disorders) | 14 | 20 | 10

LIMITATIONS AND CAVEATS:
The global study was interrupted due to issues with the clinical supply.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.